CLINICAL TRIAL: NCT03500289
Title: Ketamine for Treatment of Multiple Sclerosis-related Fatigue
Brief Title: Ketamine for Treatment of MS Fatigue
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00164017
Record Dates: First submitted 2018-04-04; First posted 2018-04-18 (Actual); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental)
  Interventions: Drug: Ketamine
- Midazolam (Placebo Comparator)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — One intravenous infusion of ketamine 0.5 mg/kg over 40 minutes
  Arms: Ketamine
Drug: Midazolam — One intravenous infusion of midazolam 0.05 mg/kg over 40 minutes
  Arms: Midazolam

SUMMARY:
Multiple sclerosis (MS) is an inflammatory, demyelinating and degenerative disease of the central nervous system and, after trauma, is the most common cause of disability in young adults, affecting more than 400,000 individuals in the US. Of all the symptoms that can occur with MS, chronic fatigue is the most common and disabling, reported by at least 75% of patients at some point. Fatigue limits patients' daily activities, and challenges employment, resulting in substantial socioeconomic consequences. Despite this negative impact, fatigue treatments have been inconsistently studied, in part due to poorly understood underlying pathophysiological mechanisms. Yet to be defined biological processes and lack of clear treatment targets have also hampered the development of drugs for fatigue. As a result, there are no medications approved by the Food and Drug Administration (FDA) for the treatment of MS fatigue.

The investigators recently reported that riluzole, a medication with anti-glutamatergic effects, increased the fatigue severity in patients with relapsing MS who had participated in a clinical trial evaluating potential neuroprotective effects of riluzole versus placebo. Three other clinic trials which examined memantine effects on cognition in patient with MS also reported worsening fatigue as a major side effect. Memantine main mechanism of action is blocking the N-methyl D-aspartate (NMDA) glutamate receptor. These observations prompted the investigators that glutamatergic transmission probably plays an important role in fatigue pathogenesis and modulating these pathways could have potential therapeutic effect on MS-related fatigue. A recent paper reported that ketamine, an NMDA receptor blocker with different kinetics compared to memantine, had a strong and prolonged effect in reducing fatigue in bipolar patients who participated in a clinical trial, evaluating anti-depressive effects of ketamine versus placebo. Interestingly, the effect of ketamine on fatigue was independent of its antidepressant effects.

The primary objective of this study is to determine if modulating glutamatergic transmission with ketamine is safe and efficacious in improving MS-related fatigue. These objectives will be answered in a proof of concept, randomized controlled trial of ketamine versus an active placebo (midazolam) in patients with relapsing or progressive MS who have clinically significant fatigue.

18 patients with MS and reported fatigue, will be randomized 2:1 to one infusion of ketamine 0.5 mg/kg over 40 minutes versus one infusion of midazolam 0.05 mg/kg over 40 minutes. Midazolam is chosen as an active placebo to keep the participants blinded to participants' medication assignment. Primary outcome of the study will be Daily Fatigue Severity measured daily from day one through day seven post-infusion.

Secondary outcomes of the study include other fatigue questionnaires, depression and sleepiness. The length of study will be around 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years 65 years.
* Females of childbearing age must have a negative urine pregnancy test at baseline and use an effective method of contraception during the study.
* Diagnosis of MS (according to the 2010 McDonald criteria).
* Ambulatory (at least 20 feet using bilateral assistance).
* Fatigue reportedly present and screening modified fatigue impact scale (MFIS) score >33.
* Internet and email access and able to use a computer or tablet

Exclusion Criteria:

* Beck Depression Inventory (BDI) score of more than 30.
* Neurodegenerative disorders other than relapsing or progressive MS.
* Breastfeeding or pregnant.
* History of coronary artery disease or congestive heart failure.
* Uncontrolled hypertension at screening (history of high blood pressure and screening systolic blood pressure >160 or diastolic blood pressure>100).
* History of severe liver disease, including cirrhosis.
* Terminal medical conditions.
* Currently treated for active malignancy.
* Alcohol or substance abuse in the past year (except marijuana or other cannabinoids).
* A history of intolerance or allergic or anaphylactic reaction to ketamine or midazolam
* Clinically unstable medical or psychiatric disorders that require acute treatment as determined by the PI.
* History of severe or untreated coronary artery disease or history of congestive heart failure.
* History of prior ischemic or hemorrhagic stroke and cerebral vascular aneurysms.
* History of recurrent seizures or epilepsy.
* Taking any disallowed therapy(ies) as noted in Appendix 2 of the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bardia Nourbakhsh, MD, MAS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Midazolam
Started | 12 | 6
Completed | 12 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Midazolam | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12.4) | 49 (8.4) | 45.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 5 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Daily Fatigue Severity Score
Description: It is a single item question: 'how much fatigue (tiredness, weariness, problems thinking clearly) have you felt today?' with responses from 0 'None at all' to 10 'Extreme Fatigue'. Reported score changes are the average point/day score change. The mean score is reported based on this calculation: [(last day measure - baseline measure) / the number of days in the study].
Time Frame: Baseline (infusion visit) through day 7
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 6
score on a scale | -0.05 [-0.19 to 0.08] | -0.05 [-0.14 to 0.24]

2. Secondary Outcome: Change in Quality of Life in Neurological Disorders (NeuroQol) Fatigue Item Bank Score
Description: T-score distributions rescale raw scores into standardized scores with a mean of 50 and a standard deviation (SD) of 10. Higher T-scores denote more severe fatigue. Reported score changes are the average point/day score change. The mean score is reported based on this calculation: [(last day measure - baseline measure) / the number of days in the study].
Time Frame: Baseline (infusion visit) through day 28 post-infusion
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 6
score on a scale | -1.02 [-1.54 to -0.5] | -0.46 [-1.20 to 0.27]

3. Secondary Outcome: Change in Modified Fatigue Impact Scale (MFIS) Score
Description: The total score of the MFIS ranges from 0 to 84. Higher scores denote more severe fatigue. Reported score changes are the average point/day score change. The mean score is reported based on this calculation: [(last day measure - baseline measure) / the number of days in the study].
Time Frame: Baseline (infusion visit) through Day 28 post-infusion
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 6
score on a scale | -0.46 [-0.70 to -0.23] | 0.02 [-0.35 to 0.32]

4. Secondary Outcome: Change in Epworth Sleepiness Scale Score
Description: The Epworth Sleepiness Scale score can range from 0 to 24. The higher the score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'. Reported score changes are the average point/day score change. The mean score is reported based on this calculation: [(last day measure - baseline measure) / the number of days in the study].
Time Frame: Baseline (infusion visit) through day 28 post-infusion
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 6
score on a scale | 0.03 [-0.18 to 0.12] | 0.11 [-0.11 to 0.32]

5. Secondary Outcome: Change in Beck Depression Inventory (BDI) Score
Description: The total score of the BDI ranges from 0 to 63. Higher scores denote more severe depressive symptoms. Reported score changes are the average point/day score change. The mean score is reported based on this calculation: [(last day measure - baseline measure) / the number of days in the study].
Time Frame: Baseline (infusion visit) through day 28 post-infusion
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 6
score on a scale | 0.07 [-0.25 to 0.11] | 0.07 [-0.33 to 0.18]

6. Secondary Outcome: Change in Fatigue Severity Scale (FSS) Score
Description: The total score of the FSS ranges from 9 to 63. Higher scores denote more severe fatigue. Reported score changes are the average point/day score change. The mean score is reported based on this calculation: [(last day measure - baseline measure) / the number of days in the study].
Time Frame: Baseline (infusion visit) through day 28 post-infusion
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 12 | 6
score on a scale | 0.03 [-0.18 to 0.12] | 0.22 [-0.11 to 0.32]

ADVERSE EVENTS:
Time Frame: One week
Arm/Group | Ketamine | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 7/12 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=12) | Midazolam (N=6)
Euphoria (Psychiatric disorders) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03500289/Prot_SAP_001.pdf